CLINICAL TRIAL: NCT00699985
Title: Comparison of Psychological Symptoms in Patients With Behcet's Disease and Control Patients by Symptom Check List 90-Revised (SCL-90-R)
Brief Title: Psychological Symptoms in Patients With Behcet's Disease by SCL90-R
Acronym: SCL90-R
Status: Completed | Type: Observational
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Rheumatology Research Center, Bahar Sadeghi
Other Study IDs: 132/11872
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Behcet's Syndrome
Keywords: Psychological Symptoms; Behcet's Disease
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Behcet's Disease patients that their diagnosis was based on the new International Criteria for Behcet's Disease (ICBD).
- 2: Non-Behcet's Disease patients were patients mimicking BD.

SUMMARY:
To find the overall psychological profile of patients with Behcet's Disease (BD) and compare it with Non-BD patients.patients were checked for psychological symptoms by Symptom Check List 90 Revised (SCL90-R)

DETAILED DESCRIPTION:
200 BD and 200 Non-BD patients were checked for psychological symptoms by Symptom Check List 90 Revised (SCL90-R). BD diagnosis was based on the new International Criteria for Behcet's Disease (ICBD). Non-BD patients were patients mimicking BD. All patients were asked to complete the SCL90-R when they attended the clinic for their routine follow-up. The demographic information and disease manifestations including ocular and neurological involvement were registered. For those with visual impairment, SCL90-R was applied by an interviewer. Frequencies and descriptive analysis were measured in both BD and Non-BD groups. Means and standard deviations (SD) of visual acuity were calculated. Data collected from SCL90-R did not have normal distribution in any dimension. The mean values of raw numbers, global severity index (GSI), the positive symptoms total (PST) and the positive symptom distress index (PSDI), were compared by Mann-Whitney U (M-W U) test.).To detect any bias in results due to data collection method, self reported data and reviewer collected data were compared.

ELIGIBILITY:
Inclusion Criteria:

* Behcet's disease patients that their diagnosis was based on the new International Criteria for Behcet's Disease (ICBD).
* Non-Behcet's disease patients were patients mimicking BD.

Exclusion Criteria:

* Probable Behcet's Disease

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: BD and Non-BD patients who attended the clinic for their routine follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2006-09; Study Completion 2007-12 (Actual)

SECONDARY OUTCOMES:
Total score of SCL90-R dimensions and global indexes | 22months

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Sadeghi, MD, Study Director — Rheumatology Research Center, Tehran University for Medical Sciences; Fereydoun Davatchi, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences; Maryam Noroozian, MD, Principal Investigator — Memory and Behavioral Department, Roozbeh Hospital, Tehran University for Medical Sciences; Farhad Shahram, MD, Principal Investigator — Rheumatology Research Center, Tehran University for Medical Sciences
Locations (1):
- Rheumatology Research Center, Shariati Hospital, Tehran, Tehran Province, Iran